CLINICAL TRIAL: NCT03451396
Title: Effect of Lifitegrast on Dry Eye Disease Signs and Symptoms
Acronym: Lifitegrast
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lifelong Vision Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5720
Record Dates: First submitted 2016-12-01; First posted 2018-03-01 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Dry Eye
Keywords: Dry eye; Tear osmolarity; Lifitegrast
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mild Dry Eye Cohort (Active Comparator): Prospective 3 month study of subjects with Tear Osmolarity >308 and VAS eye dryness ≥ 40 using 5% Lifitegrast ophthalmic solution BID.
  Interventions: Drug: Lifitegrast
- Moderate to Severe Dry Eye Cohort (Active Comparator): Prospective 3 month study of subjects with Tear Osmolarity >320 and VAS eye dryness ≥ 40 using 5% Lifitegrast ophthalmic solution BID.
  Interventions: Drug: Lifitegrast

INTERVENTIONS:
Drug: Lifitegrast — All subjects meet dry eye inclusion and will be treated with Lifitegrast gtts BID

SUMMARY:
To determine whether a fall in tear osmolarity precedes improvement in symptoms and signs of dry eye in dry eye patients treated topically with 5% lifitegrast drops for 3 months.

DETAILED DESCRIPTION:
A longitudinal, single-arm, prospective study will recruit up to 30 subjects with moderate to severe dry eye disease. Subjects will be >18 years of age, diagnosed with moderate to severe dry eye (tear osmolarity > 320 mOsm/L and Visual Analog Scale (VAS) score > 40), willing to adhere to twice daily dosing (BID) and follow up visit schedule, have no history of ocular pathology / degeneration / allergy, not on any T-cell modulatory therapy, not have instilled any artificial tears within 2 hours of study visit, and not participating in any concurrent clinical trials. All subjects will complete an informed consent form indicating their voluntary participation in the study.

Study measurements will be made at baseline (first clinic visit), 2-, 6-, and 12-weeks following Lifitegrast therapy and include tear osmolarity (TearLab osmolarity system), VAS questionnaire, slit lamp examination for fluorescein corneal staining, tear break up time (TBUT), and Meibomian gland dysfunction (MGD) grading . At the end of the 3-mo study visit, the subjects will be informed of study completion and exited from the study.

ELIGIBILITY:
Inclusion Criteria:

* Tear Osmolarity > 320 mOsm/L
* VAS eye dryness > 40
* No other ocular pathology
* No contact lens wear
* Not currently on T cell modulator
* No change in therapy in last 2 months
* Willingness to adhere to therapy and study visits
* Patients qualified for prescription of lifitegrast drops

Exclusion Criteria:

* Contact lens use
* Eye surgery in Past 6 months
* Use of tear supplements in past 2 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Primary: Tear osmolarity | Baseline to the study completion, up to 3 months.
  Number of participants with an improvement in Tear Osmolarity measured using the Tear Osmolarity score treated with Lifitegrast.

SECONDARY OUTCOMES:
VAS | VAS dry eye questionnaire, tear break up time and meibomian gland grading will be serially measured over 3 months during treatment with Lifitegrast gtts
  Participants self scored mean average on a scale of 0: none to 10: severe of Eye Dryness, Burning/Stinging, Foreign Body Sensation, Pain, Photophobia, Itching, and Blurred Vision.
Corneal Staining Grade | Baseline to the study completion, up to 3 months.
  Percentage of cornea with cell loss/fluorescein dye uptake. The higher the percentage the higher the grade.
TBUT | Baseline to the study completion, up to 3 months.
  Tear Film Break-Up Time; measurement of seconds it take for the tear film to start evaporating from the cornea.
MGD grade | Baseline to the study completion, up to 3 months.
  Visual grading of Meibomian gland clogging.

CONTACTS AND LOCATIONS:
Overall Officials: Jay S Pepose, MD, PhD, Principal Investigator — Pepose Vision Institute
Locations (1):
- Lifelong Vision Foundation, Chesterfield, Missouri, United States

REFERENCES:
- [Result] Holland EJ, Whitley WO, Sall K, Lane SS, Raychaudhuri A, Zhang SY, Shojaei A. Lifitegrast clinical efficacy for treatment of signs and symptoms of dry eye disease across three randomized controlled trials. Curr Med Res Opin. 2016 Oct;32(10):1759-1765. doi: 10.1080/03007995.2016.1210107. Epub 2016 Jul 22. PMID 27388660
- [Result] Donnenfeld ED, Karpecki PM, Majmudar PA, Nichols KK, Raychaudhuri A, Roy M, Semba CP. Safety of Lifitegrast Ophthalmic Solution 5.0% in Patients With Dry Eye Disease: A 1-Year, Multicenter, Randomized, Placebo-Controlled Study. Cornea. 2016 Jun;35(6):741-8. doi: 10.1097/ICO.0000000000000803. PMID 27055211
- [Result] Sullivan BD, Crews LA, Sonmez B, de la Paz MF, Comert E, Charoenrook V, de Araujo AL, Pepose JS, Berg MS, Kosheleff VP, Lemp MA. Clinical utility of objective tests for dry eye disease: variability over time and implications for clinical trials and disease management. Cornea. 2012 Sep;31(9):1000-8. doi: 10.1097/ICO.0b013e318242fd60. PMID 22475641